CLINICAL TRIAL: NCT06140342
Title: A Music-Based Mobile App to Combat Neuropsychiatric Symptoms in People Living With ADRD
Brief Title: A Music-Based Mobile App for People Living With Alzheimer's Disease and Related Dementias (ADRD)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Autotune Me LLC (Other)
Collaborators: University of Pennsylvania (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 3-P30-AG-073105-02 SUPPLEMENT; 3P30AG073105-02 (NIH)
Record Dates: First submitted 2023-11-03; First posted 2023-11-20 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Dementia; Agitation; Depressive Symptoms
MeSH Terms: conditions — Dementia; Psychomotor Agitation; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Feasibility study of music-based mobile app — To determine the performance and usability of the app, 20 dyads will be recruited to test it for 2 weeks. The investigators will collect physiological measures based on the application's demonstration to auto-play music according to movement or sedentary states.

SUMMARY:
The purpose of this pilot is to develop a mobile application that detects physiological measures of individuals with Alzheimer's disease and related dementias and triggers auto-play of personalized songs in a wearable device. The investigators will test the feasibility and acceptability of the app. This app may be an important tool to include in daily caregiving in a home setting by extending established benefits of music therapy for people with Alzheimer's disease and related dementias.

ELIGIBILITY:
Inclusion Criteria for person with dementia

* A person with ADRD exhibits neuropsychiatric symptoms of dementia such as agitation, restlessness, depressed mood, etc.
* Stability with or without psychotropic or anti-depressant medications
* Ability to hear with or without an assistive device

Inclusion Criteria for Caregivers

* Family or close friend caregiver of persons with dementia
* Must be able to read and write in basic English

Exclusion Criteria for all participants

* Inadequate hearing
* History of psychosis or other mental disorders other than depression
* Presence of substance or alcohol abuse

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Older adults 65+.with dementia who demonstrates symptoms of dementia such as agitation or depressive symptoms.
  Caregiver of a person with dementia
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Usability of mobile app | 2 weeks
  Dyads of caregivers of people with dementia and their caregivers will wear a smartwatch and test the music-based mobile app for two weeks. The person with dementia will wear the smartwatch that will connect to the mobile app for 2 weeks. Caregivers will be asked to complete a daily checklist of their care recipients' behaviors for two weeks.
  Participants will complete the Usefulness, Satisfaction and Ease of Use questionnaire that describes the usability of the mobile app. The minimum score is 30 while the maximum score is 240. The higher the score means the usability of the app is more acceptable.

CONTACTS AND LOCATIONS:
Locations (1):
- Autotune Me, LLC, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided